CLINICAL TRIAL: NCT01563107
Title: Dietary Sodium's Effect on Urinary Sodium and Dopamine Excretion in Patients With Postural Tachycardia Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alfredo Gamboa, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: VUMC 111633; R01HL071784 (NIH)
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Results first posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2021-12

CONDITIONS: Postural Orthostatic Tachycardia Syndrome
Keywords: Orthostatic Intolerance; Tachycardia; Orthostatic Hypotension; Sodium
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Orthostatic Intolerance; Tachycardia; Hypotension, Orthostatic | interventions — Plasma Volume

STUDY DESIGN:
Intervention Model Description: Randomization tables will be used to determine whether the 10 milliequivalents (mEq) sodium/day or 300 mEq sodium/day diet will be consumed first. Both diets will be completed on each subject (randomized crossover study), so all of the study procedures (after screening) will be repeated.
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Salt Diet (Experimental): POTS and healthy controls will be randomly assigned the order of dietary sodium levels. All procedures are performed at both levels. The high sodium diet will provide 300 milliequivalents (mEq) sodium/day.
  Interventions: Radiation: Plasma Volume; Procedure: Exercise Capacity Test - Bicycle; Procedure: Posture Study
- Low Salt Diet (Experimental): POTS and healthy controls will be randomly assigned the order of dietary sodium levels. All procedures are performed at both levels. The low sodium diet will provide 10 mEq sodium/day.
  Interventions: Radiation: Plasma Volume; Procedure: Exercise Capacity Test - Bicycle; Procedure: Posture Study

INTERVENTIONS:
Radiation: Plasma Volume — Using injection of iodinated I-131 tagged human serum albumin nominally 25 micro-Ci of radiation, blood samples are drawn before and 30 minutes after injection.
  Other Names: DAXOR
Procedure: Exercise Capacity Test - Bicycle — subjects breathe room air through a mouthpiece and exhale the air into a tube that connects to a machine (metabolic cart) that analyzes carbon dioxide and oxygen content, which allows the investigator to calculate the amount of oxygen they are using under resting and exercise conditions.
  Other Names: VO2 Max (maximal oxygen consumption)
Procedure: Posture Study — Blood pressure and heart rate will be measured while supine and then while standing for up to 30 minutes. Blood will be drawn in each position to measure hormones that regulate blood pressure and blood volume.
  Other Names: Standing Orthostatic Challenge

SUMMARY:
Patients with Postural Tachycardia Syndrome (POTS) may not adequately expand their plasma volume in response to a high sodium diet. Mechanisms involved in the regulation of plasma volume, such as the renin-angiotensin-aldosterone system and renal dopamine (DA), may be impaired in POTS and may respond inappropriately to changes in dietary sodium. The investigators propose that the changes in urinary sodium and dopamine excretion caused by consuming low-sodium and high-sodium diets will be different between patients with POTS and healthy volunteers. The purpose of this study is to determine (1) whether changes in dietary sodium level appropriately influence sodium excretion in POTS; (2) whether changes in dietary sodium level appropriately influence DA excretion in POTS; (3) whether a high dietary sodium level appropriately expands plasma volume in POTS; and (4) whether patients with POTS have improvements in their orthostatic tachycardia and symptoms as a result of a high dietary sodium level.

DETAILED DESCRIPTION:
Study Day 1

* Start 150 mEq Na+/day diet (POTS patients as inpatients; healthy control subjects with Clinical Research Center(CRC)- provided outpatient diet); consume 1.5-2 liters of water per day
* Start a 24hour (24hr) urine collection (for sodium (Na+), potassium (K+), creatinine (Cr), fractionated catecholamines)
* Blood work

Study Days 2-5

* Continue 24hr urine collection
* Start STUDY DIET (10 mEq Na+/day or 300 mEq Na+/day in a random order) after 3 meals of 150 mEq Na+/day are complete; consume 1.5-2 liters of water per day
* On Day 5, a 24 hr Holter combined ECG monitor and BP monitor will be placed on the subjects.

Study Day 6

* Continue STUDY DIET; consume 1.5-2 liters of water per day
* Remove 24hr Holter combined ECG monitor and BP monitor from subject
* Continue 24hr urine collection (for Na+, K+, Cr, fractionated catecholamines)
* Admit to CRC in afternoon (healthy control subjects only, as POTS patients will have already been admitted). Each subject will spend the night in the CRC and remain supine
* Nothing by mouth (NPO) after midnight for study next day

Study Day 7

* Awaken early (~6am) to void (still collecting 24hr urine)
* Patient returns to bed, IV catheter inserted
* Posture Study (in morning; between 7-8am ideally)
* Blood pressure and heart rate will be measured while supine and then while standing for up to 30 minutes
* We will draw blood in each body position to measure electrolytes and hormones that regulate blood pressure and blood volume
* Subjects will rate symptoms during supine period and at end of stand using Vanderbilt Orthostatic Symptoms Score (VOSS)
* Total Blood Volume (DAXOR)- using injection of iodinated I-131 tagged human serum albumin nominally 25 micro-Ci of radiation blood samples drawn through IV catheter before injection and for ~30 minutes post-injection (total - 25 ml)
* This will be done after supine assessment, but before standing the subject up
* Exercise Capacity Test (in the afternoon) Will estimate maximal oxygen consumption (VO2 max). This test will be conducted on a stationary bicycle. Effort will be gradually increased while expired air is measured during exhaustive physical work.

All procedures are repeated at least a month later with the 2nd level of dietary salt. (Randomized to high or low salt in the first phase, the second phase is the remaining level)

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal patients with POTS and healthy volunteers, 18-50 years old, who are non-smokers and free of medications with the potential to influence blood pressure
* Patients diagnosed with postural tachycardia syndrome by the Vanderbilt Autonomic Dysfunction Center
* Patients who Increase heart rate ≥30 beats/min with position change from supine to standing (10 minutes)
* For patients, chronic symptoms consistent with POTS that are worse when upright and get better with recumbence
* Only female participants are eligible. Since 80-90% of POTS patients are female, and there can be differences in measures with the menstrual cycle, including a small number of males might introduce a significant amount of noise.
* Able and willing to provide informed consent

Exclusion Criteria:

* Smokers
* Overt cause for postural tachycardia, i.e., acute dehydration
* Significant cardiovascular, pulmonary, hepatic, or hematological disease by history or screening results
* Positive pregnancy test or breastfeeding
* Hypertension defined as BP>145/95 off medications when supine or needing antihypertensive medication
* Other factors which in the investigator's opinion would prevent the participant from completing the protocol, including poor compliance during previous studies or an unpredictable schedule
* Unable to give informed consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2012-03; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Gamboa, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Healthy Participants: 17 were enrolled and randomized. 1 withdrew due to scheduling. 1 withdrew with migraines in phase 1 (low Na+). 2 withdrew in phase 1 (high Na+): 1 unable to tolerate study diet and another had difficulty cooperating with investigators.
  Postural Tachycardia Syndrome (POTS): 21 were enrolled and randomized. 6 withdrew before baseline due to age (1), pregnancy (1), prohibited meds (3), and scheduling (1). A 7th patient withdrew during phase 1 (high Na+) due to family illness.
Groups:
- Healthy Participants-Low Na+ Then High Na+: Healthy controls were randomly assigned the order of dietary sodium (Na+) levels. After baseline labs on Day 0 and 1 day on diet with150 milliequivalent (mEq) sodium/day, participants consumed low Na+ diet (10 mEq sodium/day; LS) for 6 days followed in at least 1 month by baseline labs, 1 day of 150 mEq sodium/day and 6 days of high Na+ diet (300 mEq sodium/day; HS). All procedures were performed at both levels.
- Healthy Participants-High Na+ Then Low Na+: Healthy controls were randomly assigned the order of dietary sodium (Na+) levels. After baseline labs on Day 0, and 1 day on diet with 150 milliequivalents (mEq) sodium/day,participants consumed high Na+ diet (300 mEq sodium/day; HS) for 6 days followed in at least 1 month by baseline labs, 1 day of 150 mEq sodium/day and 6 days of low Na+ diet (10 mEq sodium/day; LS). All procedures were performed at both levels.
- Patients With POTS-Low Na+ Then High Na+: Patients with POTS were randomly assigned the order of dietary sodium (Na+) levels. After baseline labs on Day 0 and 1 day on diet with 150 mEq sodium/day, participants consumed low Na+ diet (10 mEq sodium/day; LS) for 6 days followed in at least 1 month by baseline labs,1 day of 150 mEq sodium/day and 6 days of high Na+ diet (300 mEq sodium/day; HS). All procedures were performed at both levels.
- Patients With POTS-High Na+ Then Low Na+: Patients with POTS were randomly assigned the order of dietary sodium (Na+) levels. After baseline labs on Day 0 and 1 day on diet with150 mEq sodium/day, participants consumed high Na+ diet (300 mEq sodium/day; HS) for 6 days followed in at least 1 month by baseline labs, 1 day of 150 mEq sodium/day and 6 days of low Na+ diet (10 mEq sodium/day; LS). All procedures were performed at both levels.
Period: Overall Study
Arm/Group | Healthy Participants-Low Na+ Then High Na+ | Healthy Participants-High Na+ Then Low Na+ | Patients With POTS-Low Na+ Then High Na+ | Patients With POTS-High Na+ Then Low Na+
Started | 12 (12 Healthy Controls were randomized to receive LS diet followed by HS diet) | 5 (5 Healthy Controls were randomized to receive HS diet followed by LS diet) | 10 (10 POTS patients were randomized to receive LS diet followed by HS diet) | 11 (11 POTS patients were randomized to receive HS diet followed by LS diet)
Phase 1 Baseline Labs | 12 | 4 (1 healthy control was unable to find time to schedule study) | 8 (2 patients with POTS did not discontinue medication that was prohibited by protocol.) | 7 (1 patient with POTS did not discontinue medication that was prohibited by protocol, 1 patient was unable to find time to schedule the study, 1 was noted to be too old to participate, and 1 became pregnant between enrollment and the start of phase 1.)
Phase 1-150 mEq Sodium/Day | 12 | 4 | 8 | 7
Phase 1-start Low Sodium or High Sodium Diet | 12 | 4 | 8 | 7
Phase 1-finish | 11 (1 healthy control withdrew with migraines during phase 1 (low Na+).) | 2 (2 healthy controls withdrew during phase 1 (high Na+): 1 unable to tolerate study diet and another with difficulty cooperating with investigators.) | 8 | 6 (1 patient with POTS withdrew during phase 1 due to a family illness.)
Phase 2-150 mEq Sodium/Day | 11 | 2 | 8 | 6
Phase 2-start Low Sodium or High Sodium Diet | 11 | 2 | 8 | 6
Phase 2-finish | 11 | 2 | 8 | 6
Completed | 11 | 2 | 8 | 6
Not Completed | 1 | 3 | 2 | 5
Not completed — Physician Decision | 0 | 1 | 1 | 3
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Population: 14 patients with Postural Tachycardia Syndrome (POTS) and 13 Controls underwent testing while on a High Sodium Diet and while on a Low Sodium Diet, administered in a randomly assigned order. Baseline data were collected prior to starting the first dietary phase.
Groups:
- Healthy Participants-Low Na+ Then High Na+: Healthy controls were randomly assigned the order of dietary sodium (Na+) levels. After 1 day on diet with 150 mEq sodium/day, participants consumed low Na+ diet (10 mEq sodium/day; LS) for 6 days followed in at least 1 month by 1 day of 150 mEq sodium/day and 6 days of high Na+ diet (300 mEq sodium/day; HS). All procedures were performed at both levels
- HealthyParticipants-HighNa+ Then Low Na+: Healthy controls were randomly assigned the order of dietary sodium (Na+) levels. After 1 day on diet with 150 mEq sodium/day, participants consumed high Na+ diet (300 mEq sodium/day; HS) for 6 days followed in at least 1 month by 1 day of 150 mEq sodium/day and 6 days of low Na+ diet (10 mEq sodium/day; LS). All procedures were performed at both levels
- Patients With POTS-Low Na+ Then High Na+: Patients with POTS were randomly assigned the order of dietary sodium (Na+) levels. After 1 day on diet with 150 mEq sodium/day, participants consumed low Na+ diet (10 mEq sodium/day; LS) for 6 days followed in at least 1 month by 1 day of 150 mEq sodium/day and 6 days of high Na+ diet (300 mEq sodium/day; HS). All procedures were performed at both levels
- Patients With POTS-High Na+ Then Low Na+: Patients with POTS were randomly assigned the order of dietary sodium (Na+) levels. After 1 day on diet with 150 mEq sodium/day, participants consumed high Na+ diet (300 mEq sodium/day; HS) for 6 days followed in at least 1 month by 1 day of 150 mEq sodium/day and 6 days of low Na+ diet (10 mEq sodium/day; LS). All procedures were performed at both levels
- Total: Total of all reporting groups
Arm/Group | Healthy Participants-Low Na+ Then High Na+ | HealthyParticipants-HighNa+ Then Low Na+ | Patients With POTS-Low Na+ Then High Na+ | Patients With POTS-High Na+ Then Low Na+ | Total
Number analyzed (Participants) | 11 | 2 | 8 | 6 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (6) | 35 (10) | 36 (9) | 32 (6) | 33 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 2 | 8 | 6 | 27
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 10 | 2 | 8 | 5 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 9 | 2 | 8 | 6 | 25
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 2 | 8 | 6 | 27

OUTCOME MEASURES:

1. Primary Outcome: 24hr Urinary Sodium
Description: Amount of sodium excreted in urine over 24hr ending on Day 7
Time Frame: Day 6 am - Day 7 am for each dietary sodium level
Population: 24hr urine samples ending on Day 7 were collected for 13 healthy controls and 14 patients with POTS
Measure: Median (Inter-Quartile Range); unit: milliequivalents
Groups:
- Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the low sodium diet. Urine was collected daily for a 24hr period ending at approximately 8am. These results are for the final urine collection which ended on Day 7.
- Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the high sodium diet. Urine was collected daily for a 24hr period ending at approximately 8am. These results are for the final urine collection which ended on Day 7.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet.: Patients with POTS were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the low sodium diet. Urine was collected daily for a 24hr period ending at approximately 8am. These results are for the final urine collection which ended on Day 7.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet: Patients with POTS were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the high sodium diet. Urine was collected daily for a 24hr period ending at approximately 8am. These results are for the final urine collection which ended on Day 7.
Arm/Group | Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B | Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B | Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet. | Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet
Number analyzed (Participants) | 13 | 13 | 14 | 14
milliequivalents | 16.8 [12 to 26.6] | 280 [232 to 306] | 14.7 [10.8 to 22.6] | 245 [189 to 264]

2. Primary Outcome: 24hr Urinary Dopamine
Description: Amount of dopamine excreted in urine over 24 hours ending on Day 7
Time Frame: Between Day 6 am - Day 7 am of each dietary sodium level
Population: 24hr urine samples ending on Day 7 were collected for 13 healthy controls and 14 patients with POTS
Measure: Median (Inter-Quartile Range); unit: micrograms
Arm/Group | Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B | Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B | Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet. | Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet
Number analyzed (Participants) | 13 | 13 | 14 | 14
micrograms | 223 [179 to 256] | 236 [177 to 289] | 202 [150 to 258] | 205 [171 to 229]

3. Secondary Outcome: Plasma Volume
Description: Plasma volume (PV) was determined by the indicator tracer-dilution technique, using the DAXOR Blood Volume Analyzer (BVA)-100 system (DAXOR Corporation), on Day 7 of the low sodium and high sodium dietary interventions.
Time Frame: after 7 days of each dietary sodium level
Population: No data analysis for 1 healthy control who had poor venous access on Day 7 of the high sodium diet.
Measure: Median (Inter-Quartile Range); unit: mL
Groups:
- Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the low sodium diet.
  Plasma Volume: Using injection of iodinated I-131 tagged human serum albumin, blood samples were drawn before and 30 minutes after injection on Day 7 of the diet.
- Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the high sodium diet.
  Plasma Volume: Using injection of iodinated I-131 tagged human serum albumin, blood samples were drawn before and 30 minutes after injection on Day 7 of the diet.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet.: Patients with POTS were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the low sodium diet.
  Plasma Volume: Using injection of iodinated I-131 tagged human serum albumin, blood samples were drawn before and 30 minutes after injection on Day 7 of the diet.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet: Patients with POTS were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the high sodium diet.
  Plasma Volume: Using injection of iodinated I-131 tagged human serum albumin, blood samples were drawn before and 30 minutes after injection on Day 7 of the diet.
Arm/Group | Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B | Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B | Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet. | Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet
Number analyzed (Participants) | 13 | 12 | 14 | 14
mL | 2805 [2445 to 2949] | 3032 [2620 to 3482] | 2362 [2161 to 2715] | 2633 [2468 to 2961]

4. Secondary Outcome: Magnitude of Orthostatic Tachycardia
Description: Whether the magnitude of the heart rate increase that occurs in patients with POTS when moving from a supine to an upright position is attenuated by a High Sodium diet relative to a Low Sodium diet.
  Heart rate was assessed after overnight rest and fasting after midnight, following at least 60 minutes of lying quietly. Heart rate was then measured at intervals after subjects had been standing for up to 30 minutes (as tolerated). Differences between supine and standing values are presented for 5 minutes standing (or maximal stand if <5 minutes) since several patients were unable to stand for 10 minutes.
  Data in POTS patients were compared to that of Healthy Controls.
Time Frame: Supine and upright heart rate were measured after 6 days of each dietary sodium level
Population: Data is not included for 1 patient with POTS on a Low Sodium diet since that patient was unable to stand for even 1 minute.
Measure: Median (Inter-Quartile Range); unit: beats per minute
Groups:
- Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the low sodium diet.
  Supine and upright heart rate were measured on the 6th day of low sodium diet.
- Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the high sodium diet.
  Supine and upright heart rate were measured on the 6th day of high sodium diet.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet.: Patients with POTS were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the low sodium diet.
  Supine and upright heart rate were measured on the 6th day of low sodium diet.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet: Patients with POTS were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the high sodium diet.
  Supine and upright heart rate were measured on the 6th day of high sodium diet.
Arm/Group | Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B | Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B | Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet. | Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet
Number analyzed (Participants) | 13 | 13 | 13 | 14
beats per minute | 23 [19 to 36] | 19 [11 to 32] | 60 [55 to 64] | 46 [32 to 55]

5. Secondary Outcome: Upright Symptom Score
Description: Whether upright symptoms were improved in patients with POTS on a High Sodium diet relative to a Low Sodium diet.
  Patients were asked to report their standing symptom burden at the end of the Stand portion of the posture study, using the Vanderbilt Orthostatic Symptoms Scale (VOSS). They rated the severity of nine symptoms (palpitations, lightheadedness, mental confusion, blurred vision, shortness of breath, tremulousness, chest discomfort, headache, and nausea) on a scale ranging from a minimum of 0 (reflecting an absence of symptoms) to a maximum score of 10. The sum of the individual symptom scores was used to calculate orthostatic symptom burden for each participant. The lowest possible total score was 0, if a participant scored all 9 questions as 0, and the highest possible score was 90, if a participant scored all 9 questions as 10. Higher scores indicated worse symptoms.
Time Frame: Upright symptoms were assessed on the 6th day of low or high sodium diet.
Population: Upright symptom scores were inadvertently not obtained for the following number of participants:
  Healthy Participants on Low Sodium diet: 3 Healthy Participants on High Sodium diet: 2 Patients with POTS on Low Sodium diet: 5 Patients with POTS on High Sodium diet: 6
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the low sodium diet.
  Upright symptoms were assessed on the 6th day of low sodium diet.
- Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the high sodium diet.
  Upright symptoms were assessed on the 6th day of high sodium diet.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet.: Patients with POTS were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the low sodium diet.
  Upright symptoms were assessed on the 6th day of low sodium diet.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet: Patients with POTS were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the high sodium diet.
  Upright symptoms were assessed on the 6th day of high sodium diet.
Arm/Group | Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B | Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B | Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet. | Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet
Number analyzed (Participants) | 10 | 11 | 9 | 8
score on a scale | 1 [0 to 4] | 0 [0 to 3] | 30 [18 to 39] | 19 [10 to 26]

6. Secondary Outcome: Urinary Sodium Following Change in Dietary Sodium Days 1-2
Description: Urinary sodium excretion will be measured every 24 hours as the participant adapts from the 150 mEq Na/day diet to the 10 and 300 mEq Na/day diets.
Time Frame: 24 hour collections ending on Day 2 of each diet phase
Population: One healthy control neglected to collect urine during this time interval on low sodium diet, and a urine sample for another healthy control on high sodium diet was inadvertently not analyzed for sodium
Measure: Median (Inter-Quartile Range); unit: milliequivalents
Groups:
- Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the low sodium diet. Urine was collected daily for a 24hr period ending at approximately 8am. These results are for the urine collection which ended on Day 2.
- Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. . All procedures were performed at both levels. Results below were after the high sodium diet. Urine was collected daily for a 24hr period ending at approximately 8am. These results are for the urine collection which ended on Day 2.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet.: Patients with POTS were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the low sodium diet. Urine was collected daily for a 24hr period ending at approximately 8am. These results are for the urine collection which ended on Day 2.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet: Patients with POTS were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the high sodium diet. Urine was collected daily for a 24hr period ending at approximately 8am. These results are for the urine collection which ended on Day 2.
Arm/Group | Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B | Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B | Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet. | Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet
Number analyzed (Participants) | 12 | 12 | 14 | 14
milliequivalents | 145 [118 to 183] | 134 [96 to 178] | 143 [103 to 171] | 160 [95 to 180]

7. Secondary Outcome: Urinary Dopamine Following Change in Dietary Sodium Days1-2
Description: Urinary dopamine excretion will be measured every 24 hours as the participant adapts from the 150 mEq Na/day diet to the 10 and 300 mEq Na/day diets.
Time Frame: 24 hour collections ending on Day 2 of each dietary sodium phase
Population: One healthy control neglected to collect urine during this time interval on the low sodium diet
Measure: Median (Inter-Quartile Range); unit: micrograms
Groups:
- Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the high sodium diet. Urine was collected daily for a 24hr period ending at approximately 8am. These results are for the urine collection which ended on Day 2.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet.: Patients with POTS were randomly assigned the order of dietary sodium with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the low sodium diet. Urine was collected daily for a 24hr period ending at approximately 8am. These results are for the urine collection which ended on Day 2.
Arm/Group | Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B | Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B | Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet. | Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet
Number analyzed (Participants) | 12 | 13 | 14 | 14
micrograms | 228 [153 to 265] | 200 [141 to 256] | 207 [144 to 262] | 202 [159 to 228]

8. Secondary Outcome: Urinary Sodium Following Change in Dietary Sodium Days 2-3
Description: as for outcome 6
Time Frame: 24 hour collections ending on Day 3 of each diet phase
Population: 24hr urine samples were collected and analyzed for 13 healthy controls and 14 patients with POTS during both the low sodium and high sodium diet phases
Measure: Median (Inter-Quartile Range); unit: milliequivalents
Groups:
- Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the low sodium diet.
  Urine was collected daily for a 24hr period ending at approximately 8am.These results are for the urine collection which ended on Day 3.
- Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the high sodium diet.
  Urine was collected daily for a 24hr period ending at approximately 8am.These results are for the urine collection which ended on Day 3.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet.: Patients with POTS were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the low sodium diet.
  Urine was collected daily for a 24hr period ending at approximately 8am.These results are for the urine collection which ended on Day 3.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet: Patients with POTS were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Urine was collected daily for a 24hr period ending at approximately 8am.These results are for the urine collection which ended on Day 3.
Arm/Group | Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B | Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B | Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet. | Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet
Number analyzed (Participants) | 13 | 13 | 14 | 14
milliequivalents | 88.0 [73.1 to 97.4] | 199 [165 to 209] | 70.1 [60.2 to 84.6] | 154 [132 to 194]

9. Secondary Outcome: Urinary Sodium Following Change in Dietary Sodium Days 3-4
Description: as for outcome 6
Time Frame: 24 hour collections ending on Day 4 of each diet phase
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: milliequivalents
Groups:
- Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the low sodium diet.
  Urine was collected daily for a 24hr period ending at approximately 8am.These results are for the urine collection which ended on Day 4.
- Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the high sodium diet.
  Urine was collected daily for a 24hr period ending at approximately 8am.These results are for the urine collection which ended on Day 4.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet.: Patients with POTS were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the low sodium diet.
  Urine was collected daily for a 24hr period ending at approximately 8am.These results are for the urine collection which ended on Day 4.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet: Patients with POTS were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Urine was collected daily for a 24hr period ending at approximately 8am.These results are for the urine collection which ended on Day 4.
Arm/Group | Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B | Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B | Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet. | Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet
Number analyzed (Participants) | 13 | 13 | 14 | 14
milliequivalents | 32.7 [22.6 to 64.7] | 230 [177 to 261] | 28.9 [19.4 to 38.9] | 222 [203 to 265]

10. Secondary Outcome: Urinary Sodium Following Change in Dietary Sodium Days 4-5
Description: as for outcome 6
Time Frame: 24 hour collections ending on Day 5 of each diet phase
Population: The urine sample for 1 patient with POTS was collected during this time interval during high sodium diet but it was inadvertently not analyzed.
Measure: Median (Inter-Quartile Range); unit: milliequivalents
Groups:
- Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the low sodium diet.
  Urine was collected daily for a 24hr period ending at approximately 8am.These results are for the urine collection which ended on Day 5.
- Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the high sodium diet.
  Urine was collected daily for a 24hr period ending at approximately 8am.These results are for the urine collection which ended on Day 5.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet.: Patients with POTS were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the low sodium diet.
  Urine was collected daily for a 24hr period ending at approximately 8am.These results are for the urine collection which ended on Day 5.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet: Patients with POTS were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Urine was collected daily for a 24hr period ending at approximately 8am.These results are for the urine collection which ended on Day 5.
Arm/Group | Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B | Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B | Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet. | Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet
Number analyzed (Participants) | 13 | 13 | 14 | 13
milliequivalents | 17.3 [14.1 to 28.7] | 216 [182 to 249] | 21.6 [17.6 to 26.7] | 264 [258 to 309]

11. Secondary Outcome: Urinary Sodium Following Change in Dietary Sodium Days 5-6
Description: as for outcome 6
Time Frame: 24 hour collections ending on Day 6 of each diet phase
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: milliequivalents
Groups:
- Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the low sodium diet.
  Urine was collected daily for a 24hr period ending at approximately 8am.These results are for the urine collection which ended on Day 6.
- Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the high sodium diet.
  Urine was collected daily for a 24hr period ending at approximately 8am.These results are for the urine collection which ended on Day 6.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet.: Patients with POTS were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the low sodium diet.
  Urine was collected daily for a 24hr period ending at approximately 8am.These results are for the urine collection which ended on Day 6.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet: Patients with POTS were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Urine was collected daily for a 24hr period ending at approximately 8am.These results are for the urine collection which ended on Day 6.
Arm/Group | Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B | Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B | Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet. | Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet
Number analyzed (Participants) | 13 | 13 | 14 | 14
milliequivalents | 21.6 [14.6 to 31.6] | 260 [187 to 293] | 18.2 [11.6 to 25.8] | 242 [201 to 286]

12. Secondary Outcome: Urinary Dopamine Following Change in Dietary Sodium Days 2-3
Description: as for outcome 7
Time Frame: 24 hour collections ending on Day 3 of each dietary sodium phase
Population: The urine sample for 1 healthy control was collected during this interval of the low sodium diet phase, but the sample was inadvertently sent to the wrong lab for analysis
Measure: Median (Inter-Quartile Range); unit: micrograms
Groups:
- Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the low sodium diet. Urine was collected daily for a 24hr period ending at approximately 8am. These results are for the urine collection which ended on Day 3.
- Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the high sodium diet. Urine was collected daily for a 24hr period ending at approximately 8am. These results are for the urine collection which ended on Day 3.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet.: Patients with POTS were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the low sodium diet. Urine was collected daily for a 24hr period ending at approximately 8am. These results are for the urine collection which ended on Day 3.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet: Patients with POTS were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the high sodium diet. Urine was collected daily for a 24hr period ending at approximately 8am. These results are for the urine collection which ended on Day 3.
Arm/Group | Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B | Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B | Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet. | Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet
Number analyzed (Participants) | 12 | 13 | 14 | 14
micrograms | 183 [138 to 271] | 185 [126 to 250] | 205 [158 to 236] | 171 [144 to 226]

13. Secondary Outcome: Urinary Dopamine Following Change in Dietary Sodium Days 3-4
Description: as for outcome 7
Time Frame: 24 hour collections ending on Day 4 of each dietary sodium phase
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: micrograms
Groups:
- Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the low sodium diet. Urine was collected daily for a 24hr period ending at approximately 8am. These results are for the urine collection which ended on Day 4.
- Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the high sodium diet. Urine was collected daily for a 24hr period ending at approximately 8am. These results are for the urine collection which ended on Day 4.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet: Patients with POTS were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the low sodium diet. Urine was collected daily for a 24hr period ending at approximately 8am. These results are for the urine collection which ended on Day 4.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet.: Patients with POTS were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the high sodium diet. Urine was collected daily for a 24hr period ending at approximately 8am. These results are for the urine collection which ended on Day 4.
Arm/Group | Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B | Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B | Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet | Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet.
Number analyzed (Participants) | 12 | 13 | 14 | 14
micrograms | 222 [152 to 259] | 193 [128 to 244] | 203 [154 to 235] | 177 [136 to 211]

14. Secondary Outcome: Urinary Dopamine Following Change in Dietary Sodium Days 4-5
Description: as for outcome 7
Time Frame: 24 hour collections ending on Day 5 of each dietary sodium phase
Population: Urine was collected and analyzed for 13 healthy controls and 14 patients with POTS during this time interval of the low sodium and high sodium diets
Measure: Median (Inter-Quartile Range); unit: micrograms
Groups:
- Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the low sodium diet. Urine was collected daily for a 24hr period ending at approximately 8am. These results are for the urine collection which ended on Day 5.
- Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the high sodium diet. Urine was collected daily for a 24hr period ending at approximately 8am. These results are for the urine collection which ended on Day 5.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet.: Patients with POTS were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the low sodium diet. Urine was collected daily for a 24hr period ending at approximately 8am. These results are for the urine collection which ended on Day 5.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet: Patients with POTS were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the high sodium diet. Urine was collected daily for a 24hr period ending at approximately 8am. These results are for the urine collection which ended on Day 5.
Arm/Group | Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B | Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B | Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet. | Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet
Number analyzed (Participants) | 13 | 13 | 14 | 14
micrograms | 213 [145 to 253] | 202 [150 to 261] | 205 [145 to 257] | 214 [189 to 280]

15. Secondary Outcome: Urinary Dopamine Following Change in Dietary Sodium Days 5-6
Description: as for outcome 7
Time Frame: 24 hour collections ending on Day 6 of each dietary sodium phase
Population: as for outcome 14
Measure: Median (Inter-Quartile Range); unit: micrograms
Groups:
- Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the low sodium diet. Urine was collected daily for a 24hr period ending at approximately 8am. These results are for the urine collection which ended on Day 6.
- Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the high sodium diet. Urine was collected daily for a 24hr period ending at approximately 8am. These results are for the urine collection which ended on Day 6.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet.: Patients with POTS were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the low sodium diet. Urine was collected daily for a 24hr period ending at approximately 8am. These results are for the urine collection which ended on Day 6.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet: Patients with POTS were randomly assigned the order of dietary sodium levels with low sodium or high sodium diet starting after 1 day of 150 mEq sodium/day. All procedures were performed at both levels. Results below were after the high sodium diet. Urine was collected daily for a 24hr period ending at approximately 8am. These results are for the urine collection which ended on Day 6.
Arm/Group | Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B | Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B | Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet. | Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet
Number analyzed (Participants) | 13 | 13 | 14 | 14
micrograms | 227 [160 to 258] | 210 [169 to 263] | 211 [156 to 263] | 199 [168 to 251]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through discharge on the last day of phase 2 of the study. This would have been Day 8 if Low Sodium diet or Day 7 if High Sodium diet.
Description: Adverse event information was collected for any untoward or unfavorable medical occurence in a participant including any abnormal sign, symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research. Events were self-reported by participants.
Groups:
- Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the low sodium diet.
- Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B: Healthy controls were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the high sodium diet.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet.: Patients with POTS were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the low sodium diet.
- Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet: Patients with POTS were randomly assigned the order of dietary sodium levels. All procedures were performed at both levels. Results below were after the high sodium diet.
Arm/Group | Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B | Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B | Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet. | Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/13 | 1/13 | 0/14 | 0/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Participants Who Consumed Low Sodium Diet as Intervention A or Intervention B (N=13) | Healthy Participants Who Consumed High Sodium Diet as Intervention A or Intervention B (N=13) | Postural Tachycardia Syndrome (POTS) Participants Who Consumed Low Sodium Diet. (N=14) | Postural Tachycardia Syndrome (POTS) Participants Who Consumed High Sodium Diet (N=14)
Mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant notified the PI that a mass had been discovered on her pineal gland during a brain MRI for another research study. We do not believe that the mass is related to any study procedures undertaken as part of this research protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-02-22): https://cdn.clinicaltrials.gov/large-docs/07/NCT01563107/Prot_SAP_000.pdf